CLINICAL TRIAL: NCT03672760
Title: Inspiratory Muscle Training X CardioBreath App Effects On Vagal Modulation And Pulse Wave Velocity On Normotensive Postmenopause Women : Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training X CardioBreath App Effects On Vagal Modulation And Pulse Wave Velocity
Acronym: CardioBreath
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Cardiology
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Postmenopausal Disorder; Autonomic Imbalance; Vascular Stiffness

STUDY DESIGN:
Intervention Model Description: The participants will be randomized into 3 intervention groups as follows: IMT, IMT placebo and CardioBreath®App. The intervention will long five weeks. The exercises will be performed at home for five days/ week during 10 minute
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know about other arms. Outcome assessors will not know the arms participant belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMT PowerBreath (Active Comparator): Participants will have PowerBreath device for IMT adjusted for 30% of maximal inspiratory pressure and will perform the exercise at home for five days/week during 10 minutes for five weeks.
  An once a week meeting will provide re-adjustment of load through maximal inspiratory pressure performance
  Interventions: Device: IMT PowerBreath
- IMT PowerBreath Placebo (Placebo Comparator): Participants will have PowerBreath device for IMT with no load and will perform the exercise at home for five days/week during 10 minutes for five weeks.
  An once a week meeting will not re-adjustment the load though maximal inspiratory pressure performance will be performed
  Interventions: Device: IMT PowerBreath Placebo
- CardioBreathApp (Active Comparator): CardioBreathApp group will have the app settings of profile and spontaneous respiratory rate to determine the exercise rate of exercises, which will be performed at home for five days/week during 10 minutes for five weeks An once a week meeting will provide re-adjustment of respiratory rate to perform exercises
  Interventions: Device: CardioBreathApp

INTERVENTIONS:
Device: CardioBreathApp — Respiratory exercises performed with CardioBreathApp prescription and voice and visual guidance
  Arms: CardioBreathApp
Device: IMT PowerBreath — Inspiratory Muscle Training (IMT) performed with 30% load based on Maximal Inspiratory Pressure
  Arms: IMT PowerBreath
Device: IMT PowerBreath Placebo — Inspiratory Muscle Training (IMT) without load
  Arms: IMT PowerBreath Placebo

SUMMARY:
Existing data points to relevant beneficial effects of respiratory exercises on cardiovascular health, with special regards to decreases on arterial pressure and improves on autonomic and vascular profiles, though mechanistics of such results have not yet been cleared. Among the available ways to perform respiratory exercises, there is the highly recommended Inspiratory Muscle Training (IMT) and slow breathing exercises like Yoga pranayamas. Lately, the development of new technologies has allowed the use of Apps to perform respiratory exercises. This study will be take the just developed CardioBreath®App to validate it as a tool to perform respiratory exercises. Therefore, it will be compared to IMT on cardiac vagal modulation and pulse wave velocity on normotensive post menopause women.

DETAILED DESCRIPTION:
Menopause years represent an increasing risk for hypertension and autonomic nervous system (ANS) and vascular imbalance. Existing data point to beneficial effects of respiratory exercises either on ANS and light on therapeutic relevance of these kind of exercises on prevention and treatment of cardiovascular and pulmonary diseases. However, few data is available about the effects of respiratory exercises on both vascular function and interactions with ANS. Besides that, recommendations of slower respiratory rates are associated to healthier physical and psychological states. Among available techniques to perform breathing exercises, most referenced are Inspiratory Muscle Training (IMT) and Yoga based slow breathing (pranayamas). New technologies have allowed the development of Apps which aim to ease the possibilities of exercising breathing.

IMT uses a mouth device for pressure adjustment and presents a variety e training forms including combinations of intensity and volume through loads adjustment. It aims the enhancement of respiratory muscles strength and endurance.

CardioBreath®App has been developed by experienced physical education and yoga professional based on individual prescription of respiratory rates to workout through voice and image guidance of both posture and breathing technique. The performance might be followed through a progression map. It´s available in portuguese language for Android and Ios, has been submitted to Brazilian Trend Marks Institute (INPI) which has not shown opposition to the registration.

It´s a randomized clinical trial recruiting normotensive post menopause women. Eligible participants will be assessed by Finometer for blood pressure and heart rate variability as measures for autonomic outcomes. Data analysis of these data will be processed by CardioSeries software through Fourier fast transform (FFT) in order to generate vagal and sympathetic values. For pulse wave velocity and central arterial pressure the participants will be assessed by Complior Analyser.

The participants will be randomized into 3 intervention groups as follows: IMT, IMT placebo and CardioBreath®App. The intervention will long five weeks. The exercises will be performed at home for five days/ week during 10 minutes and will be registered by audio for whatsapp (IMT) and "Progress" graphics (CardioBreath®App) Once a week they will visit the laboratory set to adjust loads (IMT) and respiratory rates in CardioBreath®App groups, respectively.

After five weeks the participants will be re-evaluated for all outcomes described above.

Data analysis will be provided by ANOVA of two repeated measures and Bonferroni post hoc. All data will be presented in mean +- standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Follicle Stimulating Hormone (FSH)>35mui/ml
* minimum 12 months amenorrhea
* sedentary life style (less than 150 minutes per week of exercise)

Exclusion Criteria:

* Hypertension
* Diabetes
* Obesity
* Use of Betablockers
* recent cardiovascular events or surgery
* renal alterations
* respiratory and/or motor pathologies
* smoking
* BMI>29,9

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular autonomic control by heart rate variability(HRV) | 30 minutes
  High Frequency (HF) component of HRV (ms2 = squared milliseconds) as measure of vagal modulation

SECONDARY OUTCOMES:
Carotid -femoral pulse wave velocity (Complior) | 10 minutes
  Reduction of carotid -femoral pulse wave velocity (m/s)

OTHER OUTCOMES:
Respiratory rate by Pneumotrace respiratory belt | 30 minutes along with Finometer
  Respiratory rate in cycles per minute (CPM)
Diaphragm Thickness by ultrasound | 5 minutes
  Increase diaphragm thickness (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No